CLINICAL TRIAL: NCT06851169
Title: A Two-cohort, Exploratory Clinical Study of Perioperative Benmelstobart Alone or Combined with Anlotinib in Patients with Resectable PD-L1≥50% Non-small Cell Lung Cancer
Brief Title: This is a Two-cohort, Exploratory Clinical Study Assessing the Activity of Benmelstobart Alone or Combined with Anlotinib Administered Prior to Surgery in Terms of Pathological Complete Response
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shaanxi-Lung-002
Record Dates: First submitted 2025-01-08; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib) (Experimental): A total of 58 patients were enrolled in this exploratory study and randomly assigned to cohort 1 and cohort 2, with 29 patients in each group. Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 consecutive weeks and stopped for 1 week. Anlotinib was stopped 1 week before surgery. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 weeks and stopped for 1 week.
  Interventions: Drug: Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib)
- Cohort 2: Neoadjuvant therapy (benmelstobart only) (Experimental): Cohort 2: Neoadjuvant therapy (benmelstobart only, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1.
  Interventions: Drug: Cohort 2: Neoadjuvant therapy (benmelstobart only)

INTERVENTIONS:
Drug: Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib) — Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 consecutive weeks and stopped for 1 week. Anlotinib was stopped 1 week before surgery. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 weeks and stopped for 1 week.
  Arms: Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib)
Drug: Cohort 2: Neoadjuvant therapy (benmelstobart only) — Cohort 2: Neoadjuvant therapy (benmelstobart only, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1.
  Arms: Cohort 2: Neoadjuvant therapy (benmelstobart only)

SUMMARY:
A total of 58 patients were enrolled in this exploratory study and randomly assigned to cohort 1 and cohort 2, with 29 patients in each group. Cohort 1: Neoadjuvant therapy (benmelstobart combined with anlotinib, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 consecutive weeks and stopped for 1 week. Anlotinib was stopped 1 week before surgery. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart combined with anlotinib, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1; anlotinib, 12 mg, po, qd, was taken orally for 2 weeks and stopped for 1 week. Cohort 2: Neoadjuvant therapy (benmelstobart only, 3 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1. Surgery was performed 4-6 weeks after the final administration of benmelstobart as assessed by the investigator. Adjuvant therapy was evaluated by the investigator 4-6 weeks after surgery. Adjuvant therapy (benmelstobart, 12 cycles, every 21 days is a cycle) : benmelstobart, 1200mg, iv, day1.

ELIGIBILITY:
Inclusion Criteria:

* The participants voluntarily joined this study and signed an informed consent form. They demonstrated good compliance and cooperated well during the follow-up
* The participant must be aged between 18 and 75 years at the time of signing the informed consent form, regardless of gender
* The Eastern Cancer Collaboration (ECOG) physical fitness score was 0 or 1
* The histological confirmation of non-small cell lung cancer patients, with adequate sample size
* Resectable stage II-IIIB (IIIB limited to T2-3N2b) (according to AJCC 9th edition TNM staging)
* PD-L1 expression ≥50%
* The anticipated survival period is no less than 12 weeks
* Participants who have not undergone radiotherapy, chemotherapy, surgery, or targeted therapy prior to enrollment
* Patients with measurable lesions (RECIST 1.1)
* Both male and female patients of reproductive age agreed to the use of reliable contraceptive methods before entering the trial, during the study and up to 8 weeks after discontinuation of the drug
* Agreed to the collection of tumor histological specimens required for the study and their use in related studies
* Agreed to radical surgical treatment
* Patients with no surgical contraindications judged by specialists
* The subjects must possess adequate pulmonary function to undergo the anticipated lung resection surgery

The primary organ functions are normal and should meet the following criteria:

* Pulmonary ventilation function tests must demonstrate that FEV1 is ≥ 1.5 L, or that the expected FEV1 after lobectomy or pneumonectomy is ≥ 800 mL.
* The criteria for routine blood tests are as follows (no blood transfusions or blood products within the past 14 days, and no use of G-CSF or other hematopoietic growth factors for correction): Hemoglobin (HB) must be ≥ 90 g/L; Absolute Neutrophil Count (ANC) must be ≥ 1.5 × 10^9/L; Platelet count (PLT) must be ≥ 80 × 10^9/L.
* Biochemical examinations should meet the following criteria: Total Bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN; Serum Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance Rate (CCr) ≥ 60 mL/min.
* For patients who have not previously received anticoagulant therapy, Prothrombin Time International Normalized Ratio (INR) should be ≤ 1.5, and Activated Partial Thromboplastin Time (APTT) should be ≤ 1.5 times the upper limit of normal values. Patients receiving full-dose anticoagulant therapy or parenteral anticoagulation may enter clinical trials if their dosage has been stable for at least two weeks prior to enrollment and coagulation test results fall within local treatment limits.
* Women of childbearing age (ages 15-49 years) are required to undergo a urine pregnancy test within seven days prior to initiating treatment, with a negative result being mandatory.

Exclusion Criteria:

* Patients with large cell carcinoma, mixed cell lung cancer, and small cell lung cancer components
* Imaging (CT or MRI) shows that the tumor lesion is less than 5 mm away from the large blood vessels, there is a central tumor that is less than or equal to 2cm away from the bronchial tree; Or significant pulmonary cavity or necrotic tumor
* Any systemic anticancer treatment for NSCLC, These included cytotoxic drug therapy, immunodrug therapy, and investigational therapy
* Patients who had local radiotherapy for NSCLC
* Patients who had cancer other than NSCLC in the five years prior to the start of treatment in this study. Excluding cervical carcinoma in situ, cured basal cell carcinoma, and bladder epithelial tumors [including Ta and Tis]
* Patients who have previously used anlotinib and other anti-angiogenic agents
* Patients who have previously used benmelstobart, or other anti-PD-1, anti-PD-L1, anti-CTLA-1 antibodies, As well as any other antibody or drug therapy that targets T cell co-stimulation or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR, OX40, etc.)
* Allergy to any component of anlotinib or benmelstobart
* Multiple factors that affect oral medications (e.g. Inability to swallow, chronic diarrhea, and intestinal obstruction)
* Patients with any severe and/or uncontrolled disease, including: 1) patients with unsatisfactory blood pressure control (systolic ≥150 mmHg, diastolic ≥100 mmHg); 2) Have grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480ms), and ≥ grade 2 congestive heart failure (NYHA rating); 3) Abnormal coagulation function (INR>1.5 or prothrombin time (PT) >ULN+4 seconds or APTT >1.5 ULN), have a tendency to bleed or are receiving thrombolytic or anticoagulant therapy; Note: Under the premise of INR ≤ 1.5, the use of low dose heparin (adult daily dose of 0.6 thousand to 12 thousand U) or low dose aspirin (daily dose of 100 mg or less) is permitted for preventive purposes; 4) Active or uncontrolled serious infection; 5) Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy; 6) Renal failure requires hemodialysis or peritoneal dialysis; 7) Have a history of immunodeficiency, including HIV positive or suffering from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; 8) Poor diabetes control (fasting blood glucose (FBG) > 10 mmol/L); 9) Urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0g; 10) Patients who have seizures and require treatment; 11) Wounds or fractures that have not healed for a long time;
* Clinically significant hemoptysis (> 50ml daily hemoptysis) occurred within 2 weeks before enrollment; Or clinically significant bleeding symptoms or a definite tendency to bleed, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood ++ or above at baseline
* Patients with imaging evidence that the tumor has invaded important blood vessels or who are determined by the investigators to be highly likely to invade important blood vessels and cause fatal major bleeding during follow-up studies
* Patients with prior interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy, or any clinically demonstrated active interstitial lung disease
* Patients with acute arterial/venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism within 6 months
* Current peripheral neuropathy ≥CTCAE degree 2, except for trauma
* Subjects who underwent major surgery or had severe trauma, prior to enrollment, The effects of surgery or trauma have been resolved less than 14 days
* The patient is participating in another clinical study or has less than 4 weeks since the end of treatment in the previous clinical study
* A live or attenuated vaccine was administered within 30 days prior to the first administration of benmelstobart, or a live or attenuated vaccine was planned for the study period
* A known history of severe hypersensitivity to other monoclonal antibodies
* Pregnant or nursing women
* A clear history of neurological or psychiatric disorders, including epilepsy or dementia
* In the investigator's judgment, the patient may have other factors that might have forced the study to be terminated. Such as other serious diseases or serious laboratory abnormalities or associated with other factors that may affect the safety of the subject, or the family or society of the test data and sample collection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response (pCR) | 7 days after surgery
  Complete pathological response (pCR): defined as no residual tumor cells in postoperative tumor tissue specimens (including no tumor residue in lymph nodes), based on pathological response evaluation criteria]

SECONDARY OUTCOMES:
Major pathologic response rate (MPR) | 7 days after surgery
  Major pathologic response rate (MPR) as assessed/estimated by the investigator, i.e. the proportion of residual surviving tumor cells in the tumor bed in the postoperative specimen ≤10%
Objective response rate (ORR) | 7 days before surgery
  The proportion of patients who exhibit a partial response (PR) or complete response (CR) to treatment is defined as follows.
event-free survival (EFS) | up to 2 years
  The event-free survival (EFS) is defined as the duration from randomization to the occurrence of any event, which includes disease progression, postoperative recurrence, discontinuation of treatment for any reason, or death.
disease-free survival (DFS) | up to 2 years
  The disease-free survival period (DFS) refers to the duration from the initiation of randomization until either disease recurrence or death from any cause.
R0 removal rate | postoperative 6 hours
  Proportion of R0 level surgery performed.
overall survival (OS) | up to 3 years
  Overall survival (OS) refers to the duration from the initiation of randomization until death occurs for any reason.
Treatment-related adverse events evaluated according to CTCAE v5.0 | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Surgical complications evaluated according to the Clavien-Dindo classification | up to 2 years
  Number of participants with surgical complications as assessed by Clavien-Dindo